CLINICAL TRIAL: NCT00182273
Title: Treatment of Benign Paroxysmal Positional Vertigo With the Canalith Repositioning Procedure in Family Practice: A Randomized Controlled Trial
Brief Title: Canalith Repositioning Procedure for BPPV in Primary Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01-24
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Benign Paroxysmal Positional Vertigo
Keywords: Benign paroxysmal positional vertigo; Canalith repositioning maneuver; Dizziness; Primary Care
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Dizziness

INTERVENTIONS:
Procedure: Canalith repositioning maneuver (CRM)

SUMMARY:
The purpose of this study is to see whether family doctors can treat benign paroxysmal positional vertigo (BPPV), or dizziness, using a procedure in the office. The study is looking at whether the treatment procedure cures the dizziness in more patients compared to patients that receive a "sham" or placebo procedure.

DETAILED DESCRIPTION:
Many patients consult their family physicians because of dizziness. This is a disabling condition with serious consequences, especially in older people, as it may lead to falls and consequent fractures. One of the most common causes of dizziness is the so-called Benign Paroxysmal Positional Vertigo (BPPV). Patients with BPPV typically have severe vertigo provoked by a change in head position.

Benign Paroxysmal Positional Vertigo can now be accurately diagnosed, and distinguished form other dizziness producing conditions, in the physician's office and without any sophisticated diagnostics tools. Furthermore, it can be treated in the office setting by specific head positioning maneuvers (Canalith Repositioning Procedure) that are easy to learn and perform.

The Canalith Repositioning Procedure is currently almost exclusively performed in specialized settings by ear nose and throat (ENT) and Internal Medicine specialists. Its efficacy has been demonstrated in these settings. However, to-date no studies have been conducted in the primary care settings about the use and efficacy of the procedure, where the condition is first seen and assessed.

This is a randomized controlled trial to determine whether the procedure performed by family doctors cures dizziness.

ELIGIBILITY:
Inclusion Criteria:

* confirmed BPPV by positive Dix-Hallpike test

Exclusion Criteria:

* · Positive results of the Dix-Hallpike maneuver in both right and left head-hanging position;

  * Evidence of ongoing central nervous system disease (e.g., transient ischemic attack);
  * Otitis media;
  * Osteosclerosis;
  * Inability to tolerate a diagnostic Dix-Hallpike head-hanging maneuver;
  * Severe degenerative disc disease of cervical spine;
  * Severe and uncontrolled angina or hypertension

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56
Dates: Start 2002-01; Study Completion 2005-06

PRIMARY OUTCOMES:
Self-reported resolution (affirmative response to question: "Do you feel that the dizziness has completely resolved?") of vertigo and/or a negative result of the Dix-Hallpike maneuver

SECONDARY OUTCOMES:
Duration of cure, relapse rates

CONTACTS AND LOCATIONS:
Overall Officials: Juan Munoz, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Munoz JE, Miklea JT, Howard M, Springate R, Kaczorowski J. Canalith repositioning maneuver for benign paroxysmal positional vertigo: randomized controlled trial in family practice. Can Fam Physician. 2007 Jun;53(6):1049-53, 1048. PMID 17872784